CLINICAL TRIAL: NCT02073409
Title: Prospective Evaluation of a Standardized Approach to Diagnosis (PREDICT) and Treatment (PATIENCE) of Nontuberculous Mycobacteria Disease in Cystic Fibrosis
Brief Title: PREDICT Trial: PRospective Evaluation of NTM Disease In CysTic Fibrosis
Acronym: PREDICT
Status: Enrolling by invitation | Type: Observational
Sponsor: National Jewish Health (Other)
Collaborators: Cystic Fibrosis Foundation (Other); Children's Hospital Colorado (Other)
Responsible Party: Principal Investigator, Jerry A. Nick, M.D., Professor of Medicine, National Jewish Health
Other Study IDs: NTM-OB-17 (PREDICT PART A)
Record Dates: First submitted 2014-02-24; First posted 2014-02-27 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Cystic Fibrosis
Keywords: Nontuberculous Mycobacteria
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples collected may include serum, sputum, whole blood, breath, urine, and NTM isolates.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CF patients: Male and female subjects with CF age 6 years and older who have a positive sputum culture for NTM.

SUMMARY:
Isolation of nontuberculous mycobacteria (NTM) from the sputum of individuals with CF is an increasingly common finding, and the lack of an evidenced-based approach to the diagnosis of NTM disease has been identified as one of the greatest unmet needs within the CF community. Current evidence predicts that the prevalence of NTM will remain relatively high in the CF population. Approaches to NTM disease diagnosis differ widely between centers. This study is observational and follows current best practices. The study will help standardize the diagnosis and collect relevant data associated with the diagnosis of NTM disease to build a framework for future therapeutic trials.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent (and assent when applicable) obtained from participant or participant's legal representative
2. Enrolled in the CFF Patient Registry (CFF PR)
3. Be willing and able to adhere to study procedures in the context of clinical care, and other protocol requirements
4. Male or female participant ≥ 6 years of age at enrollment
5. Diagnosis of CF consistent with the 2017 CFF Guidelines
6. NTM positive for a species or sub-species in the 2 years prior to enrollment that has never been treated.
7. Willing to discontinue chronic azithromycin use for the duration of the study

Exclusion Criteria:

1. Prior or ongoing antibiotic treatment of the same NTM species or sub-species for which the patient is being considered for this study
2. History of solid organ or hematological transplantation
3. Has any other condition that, in the opinion of the Site Investigator/designee, would preclude informed consent or assent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Ages: 6 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female subjects with CF age 6 years and older who have a positive sputum culture for NTM.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-12; Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Proportion meeting the diagnosis of NTM disease | 12 months intervals following study enrollment

SECONDARY OUTCOMES:
Adherence to PREDICT protocol: number of respiratory cultures obtained per participant per year, withdrawals and major deviations from protocol | 12 months intervals following study enrollment
Incidence and prevalence of NTM species/subspecies by geographical region | 12 months intervals following study enrollment
Proportion of eligible NTM positive individuals with CF enrolling in PREDICT by site | 12 months intervals following study enrollment
Proportion of PREDICT participants with NTM disease diagnosis who enroll in Part B PATIENCE | 12 months intervals following study enrollment
Clinical parameters and outcomes (FEV1, growth parameters, CFQ-R) | 12 months intervals following study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Jerry A Nick, MD, Principal Investigator — National Jewish Health; Stacey Martiniano, MD, Principal Investigator — Children's Hospital Colorado
Locations (19):
- United States (19):
  - CFF Pediatric Program, University of Alabama, Birmingham, Alabama
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California San Diego, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - CFF Adult Program, Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital, Brigham & Women's Hospital, Boston, Massachusetts
  - CFF Pediatric Program University of Michigan, Ann Arbor, Michigan
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - CFF Pediatric Program, Columbia University, New York, New York
  - CFF Adult Program, University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - CFF Adult Program, The University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - CFF Pediatric Program Seattle Children's Hospital, Seattle, Washington
  - CFF Adult Program, University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Martiniano SL, Caceres SM, Poch K, Rysavy NM, Lovell VK, Armantrout E, Jones M, Anthony M, Keck A, Nichols DP, Vandalfsen JM, Sagel SD, Wagner B, Xie J, Weaver K, Heltshe SL, Daley CL, Davidson RM, Nick JA; Investigators of the Cystic Fibrosis NTM Consortium. Prospective evaluation of nontuberculous mycobacteria disease in cystic fibrosis: The design of the PREDICT study. J Cyst Fibros. 2024 Jan;23(1):50-57. doi: 10.1016/j.jcf.2023.08.007. Epub 2023 Sep 4. PMID 37666709